CLINICAL TRIAL: NCT06804577
Title: Effect of Peanut Ball Use ın Prımarıes on Labor Paın, Duratıon of Labor Anxıety and Maternal Satısfactıon
Brief Title: Effect of Peanut Ball Use ın Prımarıes on Labor Paın, Duratıon of Labor Anxıety and
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe FİLİZ (Other)
Collaborators: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Sponsor-Investigator, Ayşe FİLİZ, Principal Investigator, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: KahramanSIU
Record Dates: First submitted 2024-10-27; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: First Birth; Labor Pain; Anxiety; Birth Satisfaction
Keywords: peanut ball; labor pain; birth time; birth satisfaction
MeSH Terms: conditions — Labor Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parallel asigment
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: Educational with milnacipran (Experimental): IStage 1: When the cervical dilatation of the pregnant woman was 4-5 cm, DCO was applied after VAS 1 application. VAS 2 was applied 15 minutes after DKÖ 1 was applied.
  Stage 2: When the pregnant woman's cervical dilatation was 6-7 cm, VAS 3 was applied by the researcher. VAS 4 was applied 15 minutes after VAS 3 was applied.
  Stage 3: DKÖ 2 was applied when the pregnant woman's cervical dilatation was 7-8 cm.
  Stage 4: VAS 5 was applied when the pregnant woman's cervical dilatation was 8 cm and above. VAS 6 was applied 15 minutes after VAS 5 was applied.
  Stage 5: When the cervical effacement and dilation of the pregnant woman is completed and the fetal head rests on the perineum, the pregnant woman is taken to the delivery table.
  Stage 6: In the fourth stage of labor, between the second and third hours, the researcher will apply DCO and NDAMDS.
  Interventions: Other: peanut ball
- control group (No Intervention): standard care group

INTERVENTIONS:
Other: peanut ball — The experimental group will use peanut balls;
  Arms: Behavioral: Educational with milnacipran

SUMMARY:
Aim: The subject of this study is to examine the effects of using a peanut ball, one of the birthing ball types, on labor pain, delivery time, anxiety and maternal satisfaction in primiparous pregnant women who are planned to have a vaginal birth Material method:In the appointment, it was planned that there would be 54 people in each group. Pregnant women who meet the research criteria and agree to participate will be distributed to the groups by simple randomization method. The research sample is in the maternity unit at Gaziantep City Hospital (between August 2024 and December 2024) and all primiparous women who meet the inclusion criteria for the study will be included.

DETAILED DESCRIPTION:
Type of Study This study is a pretest-posttest randomized controlled, intervention and control two parallel group experimental study Place of Study It will be conducted in the delivery room of Gaziantep City Hospital. Research Universe: The research universe consists of primiparous pregnant women who are planned to have vaginal birth in the delivery room unit of Gaziantep City Hospital.

Research Sample Since the effect size regarding the labor comfort and labor satisfaction scales could not be obtained from the studies conducted, sample calculations could not be made for these scales in our study (Ersoy 2011, Gau et al 2011, Akın 2016, Akın and Saydam 2020). Therefore, it was determined that 60 pregnant women should be included in each group, assuming that the effect size would be 0.6 (medium), at a 5% Type I error level, and the study power was 90%. It was determined that a total of 120 primiparous pregnant women should be included in the study sample. During the study, there were no pregnant women in either group who had an emergency cesarean section or converted from normal birth to cesarean section.

Data Collection Tools The research data were collected using the Personal Information Form to determine the sociodemographic characteristics, obstetric characteristics and preparation characteristics for birth of the pregnant women, the Visual Analog Scale (VAS) to determine the labor pains perceived by the pregnant women, the State Anxiety Scale to measure the anxiety level of the pregnant women at the time of birth and the Maternal Satisfaction Evaluation Scale for Normal Birth for birth satisfaction.

Personal Information Form The form prepared by the researcher based on the literature included 11 questions regarding the sociodemographic characteristics of the women (age, height, weight, education level, marital status, employment status, income level perception, income level, place of residence, family structure, smoking); There are 5 questions about obstetric characteristics (gestational week, abortion-curettage history, pregnancy desire, regular prenatal care, where care is received) and 6 questions about preparation for birth (receiving childbirth preparation education, where education is received, preparation for motherhood, spousal support during pregnancy, family and friend support during pregnancy, satisfaction with pregnancy) for a total of 22 questions (Ersoy 2011, Chu et al 2017, Shirazi et al 2019, Kanedi et al 2019, Hildingsson and Rubertsson 2020, Akın and Saydam 2020).

VAS (Visual Analog Scale) The scale developed by Price et al. (1983) is used to determine the severity and level of pain in the patient. The scale defines pain as "0" no pain, "10" very severe on a 10 cm straight line. The patient is asked to mark a point on this line that corresponds to the level of pain he/she will feel. Accordingly, the marked point in centimeters is evaluated as the level of pain. On the scale, "0" indicates no pain, "2" indicates mild pain, "4" moderate pain, "6" severe pain, "8" very severe pain, and "10" unbearable pain. This scoring also shows the increase in the level of pain as the numerical value increases (Price 1983). State Anxiety Inventory (SAI) Spielberger's State Anxiety Inventory: The scale, developed by Spielberg and his colleagues in 1964 to measure the level of state anxiety of normal and abnormal individuals, was adapted to Turkish by Öner and Le Compte (1983). It is a self-assessment type scale consisting of short statements. The state anxiety inventory was developed to measure a person's anxiety at a certain moment. The state anxiety inventory, consisting of 20 items, is a scale that determines how an individual feels at a certain moment and under a certain condition. The feelings or behaviors expressed in the state anxiety inventory items are answered by marking one of the following options according to their intensity: (1) not at all, (2) a little, (3) a lot, (4) completely. There are 10 reversed statements in the inventory. These statements are items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The state anxiety score is calculated by adding 50 points to the difference between the total weighted scores of direct statements and reverse statements. The scores obtained in the state anxiety scale theoretically vary between 20 and 80 points. In the evaluation of the scale, it is accepted that those who score below 36 have no anxiety, those who score between 37-42 have mild anxiety, and those who score 42 and above have high anxiety (14) Normal Birth Maternal Satisfaction Assessment Scale (NDAMDS) NDAMDS was developed by Güngör and Beji (190). The relevant scale consists of a total of 43 items and 10 sub-dimensions. The sub-dimensions of the scale and item numbers are; perception of the health team (items 1, 2, 3, 4), care during labor (items 5, 6), comfort (items 7, 8, 9, 10), participation in decision-making and information (items 8, 11, 12, 13, 14, 15, 16, 17-32), meeting the baby (items 19, 20, 21), postpartum care (22, 23, 24,25, 26, 27), hospital room (28, 29, 30, 31), hospital facilities (items 32, 33, 34), privacy

ELIGIBILITY:
Inclusion Criteria Pregnant women with a singleton pregnancy, Term, primiparous, No condition preventing vaginal delivery, No extremity problems related to using a birth ball, Can speak and understand Turkish.

Exclusion Criteria Pregnant women with maternal and fetal complications (oligohydramnios and polyhydramnios, placenta previa, preeclampsia, premature membrane rupture, presentation anomalies, IUGR, fetal anomalies, intrauterine death, macrosomic baby, fetal distress, etc.) Elective cesarean section

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 1 hour
  A 10 cm ruler with no pain at one end and the most severe pain at the other end, the patient's own pain signs, the use of VAS should be explained very well. This is natural; patients are said to have two extreme points and to be free to remember between these points. The validity and reliability of the scale were made by Aslan (1998).
State Anxiety Scale (VAS) | 1 month
  Spielberger's State Anxiety Inventory: The scale was adapted to Turkish by Öner and Le Compte (1983) in 1964 by Spielberg and his friends in order to classify the degree of normal and abnormal situations. It is a self-assessment type scale consisting of short statements. The state anxiety inventory is available in a way that the person can use their anxiety at a certain moment, the state anxiety inventory consisting of 20 items is a scale that molds how the individual wants himself at a certain moment and under certain conditions. The emotions or behaviors expressed in the state record inventory classes are answered by marking one of the options (1) none, (2) a little, (3) a lot, (4) completely according to the degree of distribution. There are 10 reversed statements in the inventory. These statements are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. The state anxiety score is calculated by adding the total weighted scores of direct and reverse statements to 50 points. The scores obtai

SECONDARY OUTCOMES:
State Anxiety Scale (VAS) | 1 hour
  Spielberger's State Anxiety Inventory: The scale was adapted to Turkish by Öner and Le Compte (1983) in 1964 by Spielberg and his friends in order to classify the degree of normal and abnormal situations. It is a self-assessment type scale consisting of short statements. The state anxiety inventory is available in a way that the person can use their anxiety at a certain moment, the state anxiety inventory consisting of 20 items is a scale that molds how the individual wants himself at a certain moment and under certain conditions. The emotions or behaviors expressed in the state record inventory classes are answered by marking one of the options (1) none, (2) a little, (3) a lot, (4) completely according to the degree of distribution. There are 10 reversed statements in the inventory. These statements are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. The state anxiety score is calculated by adding the total weighted scores of direct and reverse statements to 50 points. The scores obtai

OTHER OUTCOMES:
Maternal Satisfaction Assessment Scale for Normal Birth (NDAMDÖ) | 1 hour
  NDAMDÖ was developed by Güngör and Beji (190). The relevant section consists of a total of 43 items and 10 sub-dimensions. The sub-dimensions and item numbers of the scale are; The sub-dimensions are "perceiving the health team (items 1, 2, 3, 4), care during labor (items 5, 6), comforting (items 7, 8, 9, 10), participating in decisions and informing (items 8, 11, 12, 13, 14, 15, 16, 17-32), meeting the baby (items 19, 20, 21), postpartum care (items 22, 23, 24,25, 26, 27), hospital room (items 28, 29, 30, 31), hospital facilities (items 32, 33, 34), privacy and treatment (items 35, 36, 37, 38), meeting plans (items 39, 40, 41, 42, 43)". The items are scored on a 5-point Likert-type scale according to agreement or disagreement with the statements (1-Disagree, 2-Partially disagree, 3-Undecided, 4-Agree and 5-Strongly initiated). The 13-item (products numbered 7, 8, 9,10, 19, 20, 21, 22, 35, 36, 38, 41, 42) are reverse-scored. In order to explain the scale score, the reverse scores are

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kahramanmaraş Sütçü İmam Universty, Çağlayanceri̇t, Kahramanmaraş
  - Kahramanmaraş Sütçü İmam Universty, Kahramanmaraş

IPD SHARING:
Plan to Share IPD: No